CLINICAL TRIAL: NCT04825886
Title: Evaluation of Effectiveness and Safety of ZotaRolimus-Eluting Coronary Stent System In Patients With Long Coronary Artery Disease; A Multicenter, Prospective, Observational Registry Study
Brief Title: Efficacy and Safety of ZotaRolimus-Eluting Coronary Stent System In Patients With Long Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Min Chul Kim, Associate Professor, Chonnam National University Hospital
Other Study IDs: CNUH-2017-319
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease
Keywords: Coronary Artery Disease; Zotarolimus-Eluting Stent; Long Coronary Artery Disease; Target lesion failure
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Zotarolimus-Eluting Stent — Percutaneous coronary intervention using zotarolimus-eluting stent

SUMMARY:
This study is to evaluation the efficacy and safety of Zotarolimus-Eluting Stent in patients with long coronary artery disease of 25 mm or longer.

DETAILED DESCRIPTION:
Study objectives:

From this observational prospective study, the efficacy and safety of Zotarolimus-Eluting Stent in patients with coronary artery disease longer than 25mm is planned to be investigated.

Background:

Long coronary artery lesions are observed in 20% of all coronary interventions, and are associated with poor clinical outcomes. Zotarolimus-Eluting Stents are a new type of stent that combines the advantages of an Endeavour Resolute stent (drug eluting stent) and Integrity stent (bare metal stent). In other words, BioLinx polymer is used which is an advantage of Endeavour Resolute stent to secure clinical efficiency through stable drug release while ensuring flexibility and excellent deliverability, which is the advantage of Integrity stent. To date, there are only few studies to evaluate the efficacy and safety of Zotarolimus-Eluting Stent in the treatment of coronary artery disease. Therefore, the investigators planned to carry out a multicenter, prospective observational study to evaluated the efficacy and safety of Zotarolimus-Eluting Stent in patients with long coronary artery disease of 25 mm or longer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years old
* Evidence of myocardial ischemia and coronary artery diameter stenosis≥ 50% and lesion length ≥ 25mm
* At least 2.5 mm diameter coronary vessel by visual estimation
* Patients treated with Zotarolimus-eluting stent

Exclusion Criteria:

* Previous coronary stent implantation
* Patients perticipated in other clinical trials of drugs or device
* Target vessel saphenous vein graft
* In-stent re-stenosis lesion
* Contraindicated to anti-platelet agents or hypersensitivity
* Past history of malignancy within 5 years
* History of anaphylaxis to contrast agent
* Pregnancy and lactation
* Life expectancy < 1-year
* End stage renal disease on dialysis

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery disease
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | Index admission to 12 months
  Composite endpoint of clinically driven target lesion revascularization, myocardial infarction or cardiac death related to target vessel

SECONDARY OUTCOMES:
All-cause death | Index admission, 1 month, 6 months, 12 months
  Cumulative incidence rate of all-cause death at each visit
Cardiac death | Index admission, 1 month, 6 months, 12 months
  Cumulative incidence rate of cardiac death at each visit
Myocardial Infarction | Index admission, 1 month, 6 months, 12 months
  Cumulative incidence rate of myocardial infarction at each visit
All-cause death or Myocardial infarction | Index admission, 1 month, 6 months, 12 months
  Cumulative incidence rate of all-cause death or myocardial infarction at each visit
Cardiac death or Myocardial infarction | Index admission, 1 month, 6 months, 12 months
  umulative incidence rate of cardiac death or myocardial infarction at each visit
Target vessel revascularization | Index admission, 1 month, 6 months, 12 months
  Cumulative incidence rate of target vessel revascularization at each visit
Target lesion revascularization | Index admission, 1 month, 6 months, 12 months
  Cumulative incidence rate of target lesion revascularization at each visit
Stent thrombosis | Index admission, 1 month, 6 months, 12 months
  Cumulative incidence rate of stent thrombosis at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Youngkeun Ahn, MD, Principal Investigator — Chonnam National University Hospital
Locations (20):
- South Korea (20):
  - Gyeongsang National University Changwon Hospital, Changwon
  - Dankook University Hospital, Cheonan
  - Konkuk University Medical Center, Chungju
  - Daegu Catholic University Hospital, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Eulji Medical Center, Daejeon
  - Kongyang Univeristy Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Chosun University Hospital, Gwangju
  - Wongkwang University Hospital, Iksan
  - Jeonbuk National University Hospital, Jeonju
  - Presbyterian Medical Center, Jeonju
  - Dong-A University Hospital, Pusan
  - Kosin University Gospel Hospital, Pusan
  - Paik Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Saint Carollo Hospital, Suncheon
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No